CLINICAL TRIAL: NCT00295919
Title: Phase I Study of Fenretinide (4-HPR, NSC 374551) Lym-X-Sorb™ (LXS) Oral Powder in Patients With Recurrent or Resistant Neuroblastoma
Brief Title: N2004-04: Fenretinide LXS in Treating Patients With Recurrent, Refractory, or Persistent Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Nant Operations Center, NANT Consortium, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000459787; P01CA081403 (NIH); N2004-04 (Other: NANT Consortium)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Ketoconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group (Experimental)
  Interventions: Drug: fenretinide lipid matrix; Drug: ketoconazole; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: fenretinide lipid matrix
Drug: ketoconazole
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fenretinide LXS, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase I trial is studying the side effects and best dose of fenretinide LXS in treating patients with recurrent, refractory, or persistent neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of fenretinide (4-HPR) Lym-X-Sorb™ (LXS) oral powder (4-HPR/LXS oral powder) in patients with recurrent, refractory, or persistent neuroblastoma.
* Define the toxicities of 4-HPR/LXS oral powder in these patients.
* Determine the plasma pharmacokinetics of 4-HPR/LXS oral powder and its metabolites in these patients.
* Determine the tolerability of the combination of ketoconazole and 4-HPR/LXS oral powder in these patients.

Secondary

* Determine the response rate in patients treated with 4-HPR/LXS oral powder.
* Determine the level of 4-HPR/LXS oral powder in normal peripheral blood mononuclear cells (PBMC) as a tumor cell surrogate tissue.
* Determine plasma levels of 4-HPR/LXS oral powder when given in combination with ketoconazole.
* Determine whether ketoconazole increases 4-HPR/LXS oral powder plasma levels.

OUTLINE: This is a dose-escalation study of fenretinide (4-HPR) Lym-X-Sorb™ (LXS) oral powder, followed by an open-label study. Patients are sequentially assigned to 1 of 2 intervention groups.

* Group I: Patients receive 4-HPR/LXS oral powder 3 times daily on days 0-6.
* Group II: Patients receive 4-HPR/LXS oral powder as in group I and oral ketoconazole once daily on days 0-6.

In both groups, treatment repeats every 21 days for at least 6 courses in the absence of disease progression or unacceptable toxicity. Patients in complete remission at study enrollment may receive up to 12 courses (9 months) of therapy.

Blood samples are collected at baseline and during courses 1, 2, and 6 for pharmacokinetic and correlative studies.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 32 patients will be accrued for the dose-escalation portion and 36 will be accrued for the open-label portion of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neuroblastoma either by histology and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamines
* High-risk disease, as evidenced by ≥ 1 of the following:

  * Recurrent/progressive disease at any time
  * Refractory disease (i.e., less than a partial response to frontline therapy)

    * No biopsy required
  * Persistent disease after at least a partial response to frontline therapy (i.e., patient has had at least a partial response to frontline therapy but still has residual disease by MIBG scan, CT scan/MRI, or bone marrow)

    * Biopsy of at least one residual site demonstrating viable neuroblastoma required
* Patients must have ≥ 1 of the following sites of disease:

  * Measurable tumor, defined as ≥ 2 cm in at least 1 dimension by MRI, CT scan, or x-ray OR ≥ 1 cm in at least 1 dimension by spiral CT scan

    * For persistent disease, a biopsy of bone and/or soft tissue site seen on CT/MRI must have been done to demonstrate viable neuroblastoma

      * If lesion was irradiated, biopsy must be done ≥ 2 weeks after radiation completed
  * MIBG scan with positive uptake at ≥ 1 site

    * For persistent disease, a biopsy of an MIBG-positive site must have been done to demonstrate viable neuroblastoma

      * If lesion was irradiated, biopsy must be done at least 2 weeks after radiation completed
  * Tumor cells on routine morphology (not by neuron-specific enolase staining only) of bilateral bone marrow aspirate and/or biopsy on one bone marrow sample
* Patients enrolled in group I may have had a prior relapse or progression, even if they have no measurable or evaluable tumor sites at time of study entry, including any of the following:

  * No tumor sites on all evaluations
  * Non-measurable tumor on MRI /CT scan and/or measurable tumor on CT/MRI that was previously irradiated
  * MIBG-avid site that was previously irradiated
* No CNS parenchymal or meningeal-based lesions

  * Skull-based tumor lesions with or without intracranial soft tissue extension allowed provided there are no neurological signs or symptoms or hydrocephalus related to the lesion

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 2 months
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)
* ANC ≥ 500/mm^3
* Platelet count ≥ 50,000/mm^3 (transfusion independent [ i.e., ≥ 1 week since last platelet transfusion])
* Creatinine ≤ 1.5 times normal for age as follows:

  * No greater than 0.8 mg/dL (for patients 5 years of age and under)
  * No greater than 1.0 mg/dL (for patients 6-10 years of age)
  * No greater than 1.2 mg/dL (for patients 11-15 years of age)
  * No greater than 1.5 mg/dL (for patients over 15 years of age)
* Ejection fraction ≥ 55% by echocardiogram or MUGA OR fractional shortening ≥ 27% by echocardiogram
* Bilirubin ≤ 1.5 times normal
* ALT and AST ≤ 3 times normal (for ALT, upper limit of normal is 45 U/L)
* Triglycerides < 300 mg/dL (fasting or random plasma test)
* Calcium < 11.6 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use 2 methods of effective contraception during and for 2 months after completion of study treatment
* Normal lung function (i.e., no dyspnea at rest or oxygen requirement)
* Seizure disorder allowed provided seizures are controlled on anticonvulsants that are not contraindicated
* No EKG abnormality severe enough to justify cardiac medications
* No skin toxicity > grade 1
* No hematuria and/or proteinuria > +1 on urinalysis
* No known allergy to soy products
* No known severe allergy or sensitivity to wheat gluten
* No known history of intolerance to ketoconazole (group II)

PRIOR CONCURRENT THERAPY:

* Fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy
* Prior CNS irradiation allowed
* Prior complete surgical resection of CNS lesions allowed provided there is no evidence of CNS lesions by MRI or CT scan at study entry
* At least 4 weeks since prior corticosteroid therapy for CNS lesions
* More than 3 weeks since prior myelosuppressive chemotherapy and/or biologics (4 weeks for nitrosoureas)
* More than 2 weeks since prior radiotherapy to the site of biopsied lesion or the only site of measurable disease
* At least 6 weeks since prior large-field radiotherapy (e.g., total body irradiation, craniospinal therapy, or radiotherapy to the whole abdomen, total lung, or more than 50% marrow space)
* At least 3 months since prior autologous stem cell transplantation
* At least 6 weeks since prior therapeutic MIBG
* More than 7 days since prior hematopoietic growth factors
* No prior allogeneic stem cell transplantation
* No prior organ transplantation
* No prior IV fenretinide (4-HPR) emulsion (other retinoids allowed)

  * Prior therapy with 3% 4-HPR Lym-X-Sorb™ (LXS) oral powder allowed provided patient is still on drug and it is not available for continued use
  * Prior NCI 4-HPR corn oil capsule allowed provided patient did not go off drug for toxicity
* No concurrent antiarrhythmia medications
* No other concurrent anticancer agents, including chemotherapy
* No concurrent immunomodulatory agents, including systemic corticosteroids
* No concurrent supplemental vitamin A, E, or ascorbic acid (vitamin C) except as contained in routine total parenteral nutrition vitamin supplements or in a single daily standard-dose oral multivitamin supplement
* No concurrent drugs suspected of causing pseudotumor cerebri, including tetracycline, nalidixic acid, nitrofurantoin, phenytoin, sulfonamides, lithium, amiodarone, or vitamin A (except as routine multivitamin supplement)
* No concurrent herbal supplements or other alternative therapy medications
* No concurrent medications that may potentially act as modulators of intracellular ceramide levels or ceramide cytotoxicity, sphingolipid transport, or p-glycoprotein (MDR1) or MRP1 drug/lipid transporters, including cyclosporine or analogue, verapamil, tamoxifen or analogue, ketoconazole (except if enrolled in group II), chlorpromazine, mifepristone, indomethacin, or sulfinpyrazone
* No concurrent medications that decrease gastric acid output (e.g., ranitidine) or increase gastric pH (e.g., Tums) (group II)
* No concurrent corticosteroids for emesis control

  * Systemic corticosteroids for asthma control allowed if minimized
  * Inhaled corticosteroids for asthma control and steroids for routine metabolic deficiency states allowed
* Concurrent palliative radiotherapy allowed only to sites not used to measure response

Ages: 0 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2005-12; Primary Completion 2014-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Day 1 of therapy to 16 days after last day of therapy
Toxicity of HPR/LXS oral powder | Day 1 of therapy to 16 days after last day of therapy
Plasma pharmacokinetics of 4-HPR/LXS oral powder and its metabolites | Day 0 of protocol therapy through Day 6 of Course 6
Tolerability of the combination of ketoconazole and 4-HPR/LXS oral powder | Day 1 of therapy to 16 days after last day of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Barry J. Maurer, MD, PhD, Study Chair — Texas Tech University Health Sciences Center
Locations (11):
- United States (11):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - University of Chicago Comer Children's Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington

REFERENCES:
- [Result] Marachelian A, Kang MH, Hwang K, et al.: Phase I study of fenretinide (4-HPR) oral powder in patients with recurrent or resistant neuroblastoma: New Approaches to Neuroblastoma Therapy (NANT) Consortium trial. [Abstract] J Clin Oncol 27 (Suppl 15): A-10009, 2009.